CLINICAL TRIAL: NCT00451295
Title: A Phase III, Double-Blind, Multi-Centre, Randomised, Parallel Group Design, Placebo-Controlled, Flexible Dose Study of MCI-196 in Combination With a Ca-Based Phosphate Binder in CKD Stage V Subjects on Dialysis With Hyperphosphatemia.
Brief Title: A Phase III, Multi-Centre, Randomised, Placebo-Controlled Study in Combination With Ca-based P Binders in Patients With Hyperphosphatemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped because of insufficient enrollment.
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCI-196-E09
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Kidney Disease; Dialysis; Hyperphosphatemia
Keywords: Chronic Kidney Disease; Dialysis; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — cholebine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: MCI-196(colestilan(INN), Colestimide(JAN), CHOLEBINE®)

INTERVENTIONS:
Drug: MCI-196(colestilan(INN), Colestimide(JAN), CHOLEBINE®) — 3g to 15g/day (3 times a day), Tablet, 12 weeks of flexible dose
  Arms: 2
Drug: Placebo — 3g to 15g/day (3 times a day), Tablet, 12 weeks of flexible dose
  Arms: 1

SUMMARY:
This study consists of a 4 week run-in period with a Ca based phosphate binder and 12 weeks treatment period by MCI-196 or placebo, (both on Ca based phosphate binder). During the treatment period, MCI-196 or placebo will be titrated every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 80 years of age.
2. Stable phosphate control using Calcium-based phosphate-binding medication only.
3. The subject is undergoing regular dialysis treatment.
4. On a stabilised phosphorus diet.
5. If female and of child-bearing potential, has a negative serum pregnancy test. Sexually active females must agree to take appropriate steps not to become pregnant.
6. Male subjects must agree to use appropriate contraception.

Exclusion Criteria:

1. Current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose them to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
2. Body mass index (BMI) <=16.0 kg/m2 or =>40.0 kg/m2.
3. Current or a history of significant gastrointestinal motility problems
4. A positive test for hepatitis B surface antigen, hepatitis C antibody or HIV 1 and 2 antibodies.
5. A history of substance or alcohol abuse within the last year.
6. Seizure disorders.
7. Using phosphate binder medication other than calcium based phosphate binders
8. Using colestyramine, colestipol or colesevelam
9. A history of drug or other allergy
10. Participated in a clinical study with any experimental medication in the last 30 days or an experimental biological product within the last 90 days, prior to signing of the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus change compared to placebo from baseline to week 12. | 12 weeks

SECONDARY OUTCOMES:
Both Efficacy parameters (such as LDL-cholesterol, other lipid parameters, PTH, Ca, Ca x P ion product) and safety parameters. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma Europe
Locations (25):
- Czechia (2):
  - Frýdek-Místek
  - Ostrava
- France (2):
  - Bordeaux
  - Montpelier
- Germany (2):
  - Aachen
  - Coburg
- Italy (3):
  - Lecco
  - Milan
  - Pavia
- Skopje, North Macedonia
- Poland (7):
  - Gdansk
  - Krakow
  - Lodz
  - Oświęcim
  - Poznan
  - Wejherowo
  - Wroclaw
- Serbia (3):
  - Belgrade
  - Niš
  - Novisad
- South Africa (2):
  - Cape Town
  - Gauteng
- Spain (2):
  - Barcelona
  - Oviedo
- Stevenage, United Kingdom